CLINICAL TRIAL: NCT00974428
Title: A 6 Week, Double Blind, Placebo-controlled, Multi-center Pilot Study Evaluating the Efficacy of Wobenzym(R)N at Reducing Pain Severity as Measured by the WOMAC Pain Score in Subjects With Knee Osteoarthritis
Brief Title: Multi-Center Study Evaluating the Efficacy of Wobenzym(R)N in Treating Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Atrium Innovations (Industry)
Responsible Party: Barry W. Ritz/Vice President for Scientific Affairs, Atrium Innovations
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A077-ATR08H
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Disease of joints; Wobenzym® N; WOMAC pain score; Subject reported pain (VAS)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Wobenzym® N and placebo (Active Comparator): Wobenzym® N 2 tablets of the treatment and 2 placebo tablets three times per day
  Interventions: Dietary Supplement: Wobenzym® N; Dietary Supplement: Placebo
- Wobenzym® N (Active Comparator): Wobenzym® N 4 tablets three times per day
  Interventions: Dietary Supplement: Wobenzym® N
- Placebo (Placebo Comparator): Placebo 4 tablets three times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wobenzym® N — 4 tablets TID, 6 weeks
  Other Names: None known.
  Arms: Wobenzym® N; Wobenzym® N and placebo
Dietary Supplement: Placebo — 4 tablets TID
  Other Names: None known.
  Arms: Placebo; Wobenzym® N and placebo

SUMMARY:
The objective of this study is to determine the most effective dose of Wobenzym® N versus placebo at reducing pain severity as measured by the WOMAC pain score in subjects with symptomatic knee osteoarthritis (OA) at 6 weeks of treatment.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common disease of the joints. The main symptom of OA is pain and later followed by stiffness and decreased function of the joints. It is estimated to affect more than 100 million people worldwide, substantially decreasing their quality of their life. Treatment that can relieve the disease symptoms and more particularly the pain level can greatly improve the quality of life and function of patients suffering from OA of weight-bearing joints such as the knee. Wobenzym® N is a fixed compound made of plant and animal enzyme products with the non-enzymatic component rutin recommended for the treatment of musculoskeletal disorders. The Wobenzym® N formulation contains, per tablet: pancreatin 100 mg, trypsin 24 mg and chymotrypsin 1 mg (from pancreas); bromelain 45 mg; papain 60 mg; and rutin 50 mg.

Over 50 clinical studies have been conducted using similar oral proteolytic enzyme preparations-- Wobenzym® and Phlogenzym®-- with consistently positive findings related to rheumatoid arthritis, sprains and strains, reduction of C-reactive protein, sports injuries and joint and muscular pain, as well as OA of the knee. Several comparative studies conducted with Phlogenzym®, an oral enzyme-rutin combination containing bromelain 90 mg, trypsin 48 mg and rutin 100 mg, have proved the product to be effective and safe in the treatment of OA as compared to NSAIDs. [For review, see Leipner, et al. Biodrugs 2001;15(12):779-89.]

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory outpatients of either sex, between 45 and 80 years of age, inclusively, with primary OA of the knee meeting the classification criteria set by the American College of Rheumatology (ACR; Appendix C.1), and who are not expected to require surgical treatment for at least three (3) months after inclusion (Visit 1).
* Women of childbearing potential must agree to use an adequate contraception (abstinence; device mechanical barrier contraception; male partner sterilized) beginning at least seven days prior to treatment (oral birth control pill should begin at least 4 weeks prior to treatment) and continuing at least 14 days after Visit 4 or the discontinuation visit. A serum or urine pregnancy test will be performed at Visit 1.
* Functional Capacity Classification (Appendix C.2) of I-III at Visit 1.
* Except for OA, the subject is judged to be in otherwise general good health based on medical history, physical examination, and routine laboratory tests (Appendix B).
* Subjects with a WOMAC pain subscale index of at least 40 mm and less than or equal to 90 mm (VAS) at the Baseline Visit after a 24-hour washout of any analgesics and a minimum of 7 days washout of any NSAIDs (Appendix C.3 & 4).
* Subjects with OA of the contra-lateral knee will be included provided contra-lateral knee OA pain intensity is inferior to the index knee.
* Able to understand and complete study questionnaires including questions requiring a visual analog scale (VAS) response (Appendix C.4).
* Willing to participate in this study for approximately ten weeks.
* Written informed consent obtained.
* Subject agreed to follow the protocol.

Exclusion Criteria:

* Any contraindication to the use of Wobenzym® N (including allergy).
* Concurrent medical/arthritic disease that could confound or interfere with the monitoring of efficacy including, but no limited to: Inflammatory arthritis (e.g., rheumatoid arthritis), systemic lupus, spondyloarthropathy, psoriatic arthropathy, Reiter's syndrome, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, polymyalgia rheumatica and gout or pseudogout of the index knee, Paget's disease affecting the study joint, a history of septic arthritis or intra-articular fracture of the study joint, osteochondritis, dessicans or osteonecrosis of the study joint, Wilson's disease, haemochromatosis, ochronosis, chondrocalcinosis or primary osteochondromatosis.
* Significant injury of the study joint within three months of the Baseline visit as per investigator judgment.
* Subjects with Class IV functional capacity using the ACR criteria.
* Subjects who had meniscal surgery on the study knee.
* Subjects who have undergone total joint replacement of the contra-lateral knee within six months prior to the Screening Visit (Visit 1).
* Any clinical signs or laboratory evidence for severe renal/liver/pulmonary, neurological, cardiovascular, metabolic, haematological, or psychiatric condition which in the Investigator's opinion contraindicates a 6 week course of therapy with Wobenzym® N.
* Subject is, in the opinion of the investigator, mentally or legally incapacitated preventing informed consent from being obtained, or cannot read or comprehend written material.
* Active malignancy of any type or history of a malignancy within the last five years other than basal cell carcinoma.
* Any active gastrointestinal disease.
* Use of NSAID within seven days of entering the study (Visit 2).
* Use of glucosamine sulphate, chondroitin sulphate or any other natural health product and/or OTC product that claim to be effective for pain and/or OA within 30 days of entering the study (Visit 2).
* History of drug abuse or active alcoholism.
* Any investigational drug within 30 days prior to screening.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Determination of the most effective dose of Wobenzym® N on the reduction of pain severity, measured by the WOMAC Osteoarthritis Index. | Baseline (day 0), Week 3 (day 21) and Week 6 (day 42)

SECONDARY OUTCOMES:
Subject Global assessment | Week 3 (day 21) and Week 6 (day 42)
Subject assessment of pain (VAS) | Baseline (day 0), Week 3 (day 21) and Week 6 (day 42)
Inflammatory profile (serum biomarkers) in serum samples | Screening visit (-30 days prior day 0) and Week 6 (day 42)

CONTACTS AND LOCATIONS:
Overall Officials: André Beaulieu, Dr, Principal Investigator — Centre de Rhymatologie St-Louis; Louis Bessette, Dr, Principal Investigator — Groupe de recherche en rhumatologie et maladies osseuses; Morin Frédéric, Dr., Principal Investigator — Centre de Recherche Musculo-Squelettique; Jean-Pierre Raynauld, Dr, Principal Investigator — Institut de rhumatologie de Montréal
Locations (4):
- Canada (4):
  - Institut de Rhumatologie de Montréal, Montreal, Quebec
  - Groupe de Recherche en Rhumatologie et maladies osseuses, Québec, Quebec
  - Centre de Rhumatologie St-Louis, Sainte-Foy, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec